CLINICAL TRIAL: NCT06939361
Title: The Tube Size Randomized Trial During Emergency Tracheal Intubation
Brief Title: Tube Size Randomized Trial During Emergency Tracheal Intubation
Acronym: BREATHE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Primary Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250125
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Failure
Keywords: critical illness; emergency airway management; tracheal intubation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Parallel-group, pragmatic, randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smaller Endotracheal Tube Group (Active Comparator): For patients assigned to the smaller endotracheal tube group, the operator will place a smaller endotracheal tube, as defined below:
  * Inner diameter 7.0 mm (for patients with a height ≥ 64 inches)
  * Inner diameter 6.5 mm (for patients with a height < 64 inches)
  Interventions: Other: Smaller endotracheal tube
- Larger Endotracheal Tube Group (Active Comparator): For patients assigned to the larger endotracheal tube group, the operator will place a larger endotracheal tube, as defined below:
  * Inner diameter 8.0 mm (for patients with a height ≥ 64 inches)
  * Inner diameter 7.5 mm (for patients with a height < 64 inches)
  Interventions: Other: Larger endotracheal tube

INTERVENTIONS:
Other: Smaller endotracheal tube — * Inner diameter 7.0 mm (for patients with a height ≥ 64 inches)
  * Inner diameter 6.5 mm (for patients with a height < 64 inches)
  Arms: Smaller Endotracheal Tube Group
Other: Larger endotracheal tube — * Inner diameter 8.0 mm (for patients with a height ≥ 64 inches)
  * Inner diameter 7.5 mm (for patients with a height < 64 inches)
  Arms: Larger Endotracheal Tube Group

SUMMARY:
The BREATHE trial is a parallel-group, pragmatic, randomized clinical trial comparing the effectiveness of smaller versus larger endotracheal tubes for mechanical ventilation of critically ill adults at 7 geographically diverse centers. A total of 3,180 critically ill adults undergoing tracheal intubation in the ED or ICU will be enrolled. Enrolled patients will be randomly assigned in a 1:1 ratio to receive either a smaller endotracheal tube (a 6.5 mm endotracheal tube for patients shorter than 64 inches and a 7.0 mm endotracheal for patients at least 64 inches) or a larger endotracheal tube (a 7.5 mm endotracheal tube for patients shorter than 64 inches and a 8.0 mm endotracheal for patients at least 64 inches). Patients will be followed for 6 months after enrollment. The primary outcome will be breathlessness at 6 months. The secondary outcomes will be voice quality and swallowing at 6 months.

DETAILED DESCRIPTION:
Each year, approximately 1% of the US population (2-3 million adults) experiences critical illness requiring placement of an endotracheal tube. While 60-80% of patients survive, more than half of survivors experience long-term problems with breathing, speaking, or swallowing. Identifying approaches that prevent long-term complications of critical illness is an urgent priority.

For every patient undergoing emergency tracheal intubation, clinicians select the size of endotracheal tube. The size of the endotracheal tube refers to the inner diameter of the tube. Smaller endotracheal tubes commonly used in adults have a diameter of 6.5 mm to 7.0 mm. Larger endotracheal tubes commonly used in adults have a diameter of 7.5 mm to 8.0 mm.

In current clinical care, some clinicians routinely use smaller endotracheal tubes while others routinely use larger endotracheal tubes. In a cohort of 2,652 patients enrolled in three recent trials conducted by our Pragmatic Critical Care Research Group (PCCRG), clinicians used a smaller endotracheal tube for 44.5% of patients and a larger endotracheal tube for 55.5%. While height and sex are the primary determinants of the diameter of a patient's trachea, these variables explain only 12% of the variation in the size of endotracheal tube clinicians use in current clinical care. This suggests that selection of endotracheal tube size in clinical practice is not "personalized" to the characteristics of the patient, but instead varies based on factors like the specialty of the clinician, the practice patterns of the hospital, and the region of the country.

Whether using a smaller vs larger endotracheal tube affects any patient outcome is unknown. Some experts have hypothesized that use of larger endotracheal tubes may cause acute injury to the larynx, which for some patients could progress to permanent scarring, impairing breathing, speaking, and swallowing. Thus, some experts currently recommend using smaller endotracheal tubes. Other experts hypothesize that the use of larger endotracheal tubes may reduce resistance to gas flow, reducing patients' work of breathing during spontaneous breathing trials, and making it easier to pass suction catheters, obtain diagnostic samples, and clear secretions. Such experts, therefore, currently recommend using larger endotracheal tubes in hopes that doing so might shorten the duration of invasive mechanical ventilation or even decrease the risk of death during critical illness. No randomized trials have ever compared smaller versus larger endotracheal tube sizes among critically ill adults. Only one observational study has evaluated the effect of endotracheal tube size on outcomes of critical illness. It suggested that smaller endotracheal tubes had no effect on survival to hospital discharge but could not exclude the possibility that endotracheal tube size might affect the duration of invasive mechanical ventilation. The study prompted published responses highlighting the lack of long-term outcomes and the biases inherent to observational studies, noting that the effects of smaller versus larger endotracheal tubes could only be proven with a randomized trial.

Because millions of critically ill adults receive either a smaller or larger endotracheal tube during tracheal intubation in an ED or ICU each year, and no prior randomized trial has evaluated the effect of endotracheal tube size on long-term outcomes (breathing, speaking, and swallowing) or short-term outcomes (duration of invasive mechanical ventilation and survival), a multicenter randomized trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing orotracheal intubation with an endotracheal tube in a participating unit
* Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit

Exclusion Criteria:

* Patient is known to be less than 18 years old
* Patient is known to be pregnant
* Patient is known to be a prisoner
* Use of an endotracheal tube with subglottic suction is planned
* Operator has determined that use of a smaller endotracheal tube or a larger endotracheal tube is required or contraindicated for the optimal care of the patient
* Immediate need for tracheal intubation precludes safe performance of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3180 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Breathlessness at 6 months after intubation | At 6 months after enrollment
  Primary Effectiveness Outcome: Breathlessness will be measured using the Clinical COPD Questionnaire (CCQ). Scores range from 0 (least severe) to 6 (most severe).

SECONDARY OUTCOMES:
Ventilator-free days in the first 28 days | From enrollment to 28 days after enrollment
  Primary Safety Outcome: The number of days alive and free of invasive mechanical ventilation from enrollment to 28 days after enrollment.
All-cause, in-hospital mortality by 28 days | From enrollment to 28 days after enrollment
  Primary Safety Outcome: Death from any cause from enrollment to 28 days after enrollment, censored at hospital discharge.
Voice impairment at 6 months after intubation | At 6 months after enrollment
  Secondary Effectiveness Outcome: voice impairment at 6 months after enrollment as measured using the Voice Handicap Index (VHI) survey. Scores range from 0 (least severe) to 40 (most severe).
Swallowing impairment at 6 months after intubation | At 6 months after enrollment
  Secondary Effectiveness Outcome: Swallowing impairment at 6 months after enrollmnet as measured using the EAT-10 survey. Scores range from 0 (least severe) to 40 (most severe).

OTHER OUTCOMES:
Successful intubation on the first attempt. | Duration of placement of the endotracheal tube, an average duration of two minutes
  Successful intubation on the first attempt is defined as placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and EITHER a single insertion of an endotracheal tube into the mouth OR a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube over the bougie into the mouth.
Number of laryngoscopy attempts | Duration of placement of the endotracheal tube, an average duration of two minutes
Number of attempts to cannulate the trachea with a bougie | Duration of placement of the endotracheal tube, an average duration of two minutes
Number of attempts to cannulate the trachea with an endotracheal tube | Duration of placement of the endotracheal tube, an average duration of two minutes
Time from initiation of laryngoscopy to intubation of the trachea | Duration of placement of the endotracheal tube, an average of 60 seconds
  Time from initiation of laryngoscopy to intubation of the trachea in seconds
Severe hypoxemia | During procedure (between induction and 2 minutes after tracheal intubation).
  Lowest oxygen saturation <80%
Agitation | From intubation to 7 days after enrollment
  As measured by the occurrence of a Richmond Agitation-Sedation Scale (RASS) ≥ +2
Delirium | From intubation to 7 days after enrollment
  As measured by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
Tracheostomy | From intubation to 28 days after enrollment
  Occurence of a tracheostomy procedure.
Percutaneous gastrostomy tube placement | From intubation to 28 days after enrollment
  Occurence of a gastrostomy tube placement.
Endotracheal tube exchange | From intubation to 28 days after enrollment
  Exchange of the endotracheal tube for any reason during the index course of invasive mechanical ventilation
Reintubation within 72 hours of extubation from the index course of invasive mechanical ventilation | Within 72 hours of extubation
  Any placement of an endotracheal tube in the trachea (e.g., endotracheal tube, tracheostomy) between extubation from the index course of invasive mechanical ventilation and 72 hours following extubation, excluding reintubations for the purpose of a procedure that lasts <24 hours.
Ventilator associated pneumonia during the index course of invasive mechanical ventilation | From intubation to 28 days after enrollment
  New lung infiltrate plus clinical evidence that the infiltrate is of an infectious origin, which include the new onset of fever, purulent sputum, leukocytosis, and decline in oxygenation, beginning > 48 hours after enrollment.
ICU-free days in the 28 days after enrollment | From intubation to 28 days after enrollment
Hospital-free days in the 28 days after enrollment | From intubation to 28 days after enrollment
All-location mortality by 28 days | At 28 days after enrollment
All-cause, all-location mortality by 6 months | At 6 months after enrollment
Prescence of a tracheostomy at 6 months | At 6 months after enrollment
Cough at 6 months | At 6 months after enrollment
  As measured by the Cough Severity Index. Scores range from 0 (no cough) to 40 (severe cough).
Throat pain at 6 months | At 6 months after enrollment
  As measured by the Numeric Rating Scale. Scores range from 0 (no pain) to 10 (most severe pain).
Voice quality at 6 months | At 6 months after enrollment
  As measured by the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V). Scores range from 0 (mildly deviant) to 100 (severely deviant).
Quality of life at 6 months | At 6 months after enrollment
  As measured by the EQ-5D-5L health-related quality of life measure. Scores range from 0 (worst health) to 100 (best health).
Anxiety at 6 months | At 6 months after enrollment
  As measured by the General Anxiety Disorder-7 (GAD-7). Scores range from 0 (least severe) to 21 (most severe).
Depression at 6 months | At 6 months after enrollment
  As measured by the Patient Health Questionnaire-9. Scores range from 0 (not at all) to 27 (nearly every day).
Employment at 6 months | At 6 months after enrollment
  As measured by the OACIS Employment Questionnaire.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of Colorado-Denver, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Kempker JA, Abril MK, Chen Y, Kramer MR, Waller LA, Martin GS. The Epidemiology of Respiratory Failure in the United States 2002-2017: A Serial Cross-Sectional Study. Crit Care Explor. 2020 Jun 10;2(6):e0128. doi: 10.1097/CCE.0000000000000128. eCollection 2020 Jun. PMID 32695994
- [Background] Heidegger T. Management of the Difficult Airway. N Engl J Med. 2021 May 13;384(19):1836-1847. doi: 10.1056/NEJMra1916801. No abstract available. PMID 33979490
- [Background] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Background] Driver BE, Prekker ME, Moore JC, Schick AL, Reardon RF, Miner JR. Direct Versus Video Laryngoscopy Using the C-MAC for Tracheal Intubation in the Emergency Department, a Randomized Controlled Trial. Acad Emerg Med. 2016 Apr;23(4):433-9. doi: 10.1111/acem.12933. Epub 2016 Mar 24. PMID 26850232
- [Background] Demoule A, Hajage D, Messika J, Jaber S, Diallo H, Coutrot M, Kouatchet A, Azoulay E, Fartoukh M, Hraiech S, Beuret P, Darmon M, Decavele M, Ricard JD, Chanques G, Mercat A, Schmidt M, Similowski T; REVA Network (Research Network in Mechanical Ventilation). Prevalence, Intensity, and Clinical Impact of Dyspnea in Critically Ill Patients Receiving Invasive Ventilation. Am J Respir Crit Care Med. 2022 Apr 15;205(8):917-926. doi: 10.1164/rccm.202108-1857OC. PMID 35061577
- [Background] Nanwani-Nanwani K, Lopez-Perez L, Gimenez-Esparza C, Ruiz-Barranco I, Carrillo E, Arellano MS, Diaz-Diaz D, Hurtado B, Garcia-Munoz A, Relucio MA, Quintana-Diaz M, Urbez MR, Saravia A, Bonan MV, Garcia-Rio F, Testillano ML, Villar J, Garcia de Lorenzo A, Anon JM. Prevalence of post-intensive care syndrome in mechanically ventilated patients with COVID-19. Sci Rep. 2022 May 13;12(1):7977. doi: 10.1038/s41598-022-11929-8. PMID 35562379
- [Background] Dowdy DW, Eid MP, Dennison CR, Mendez-Tellez PA, Herridge MS, Guallar E, Pronovost PJ, Needham DM. Quality of life after acute respiratory distress syndrome: a meta-analysis. Intensive Care Med. 2006 Aug;32(8):1115-24. doi: 10.1007/s00134-006-0217-3. Epub 2006 Jun 17. PMID 16783553
- [Background] Heyland DK, Groll D, Caeser M. Survivors of acute respiratory distress syndrome: relationship between pulmonary dysfunction and long-term health-related quality of life. Crit Care Med. 2005 Jul;33(7):1549-56. doi: 10.1097/01.ccm.0000168609.98847.50. PMID 16003061
- [Background] Hudson LD. What happens to survivors of the adult respiratory distress syndrome? Chest. 1994 Mar;105(3 Suppl):123S-126S. doi: 10.1378/chest.105.3_supplement.123s. No abstract available. PMID 8131606
- [Background] Davidson TA, Caldwell ES, Curtis JR, Hudson LD, Steinberg KP. Reduced quality of life in survivors of acute respiratory distress syndrome compared with critically ill control patients. JAMA. 1999 Jan 27;281(4):354-60. doi: 10.1001/jama.281.4.354. PMID 9929089
- [Background] Miles A, McRae J, Clunie G, Gillivan-Murphy P, Inamoto Y, Kalf H, Pillay M, Pownall S, Ratcliffe P, Richard T, Robinson U, Wallace S, Brodsky MB. An International Commentary on Dysphagia and Dysphonia During the COVID-19 Pandemic. Dysphagia. 2022 Dec;37(6):1349-1374. doi: 10.1007/s00455-021-10396-z. Epub 2022 Jan 4. PMID 34981255
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Brodsky MB, Gonzalez-Fernandez M, Mendez-Tellez PA, Shanholtz C, Palmer JB, Needham DM. Factors associated with swallowing assessment after oral endotracheal intubation and mechanical ventilation for acute lung injury. Ann Am Thorac Soc. 2014 Dec;11(10):1545-52. doi: 10.1513/AnnalsATS.201406-274OC. PMID 25387319
- [Background] Karmali S, Rose P. Tracheal tube size in adults undergoing elective surgery - a narrative review. Anaesthesia. 2020 Nov;75(11):1529-1539. doi: 10.1111/anae.15041. Epub 2020 May 16. PMID 32415788
- [Background] Karmakar A, Pate MB, Solowski NL, Postma GN, Weinberger PM. Tracheal size variability is associated with sex: implications for endotracheal tube selection. Ann Otol Rhinol Laryngol. 2015 Feb;124(2):132-6. doi: 10.1177/0003489414549154. Epub 2014 Oct 10. PMID 25305266
- [Background] Dominelli PB, Ripoll JG, Cross TJ, Baker SE, Wiggins CC, Welch BT, Joyner MJ. Sex differences in large conducting airway anatomy. J Appl Physiol (1985). 2018 Sep 1;125(3):960-965. doi: 10.1152/japplphysiol.00440.2018. Epub 2018 Jul 19. PMID 30024341
- [Background] Eckel HE, Sittel C. Morphometry of the larynx in horizontal sections. Am J Otolaryngol. 1995 Jan-Feb;16(1):40-8. doi: 10.1016/0196-0709(95)90008-x. PMID 7717472
- [Background] Mir F, Sandhu G, Poncia J. Size matters: choosing the right tracheal tube. Anaesthesia. 2012 Dec;67(12):1402-3; author reply 1403-4. doi: 10.1111/anae.12026. No abstract available. PMID 23130729
- [Background] Gelbard A, Francis DO, Sandulache VC, Simmons JC, Donovan DT, Ongkasuwan J. Causes and consequences of adult laryngotracheal stenosis. Laryngoscope. 2015 May;125(5):1137-43. doi: 10.1002/lary.24956. Epub 2014 Oct 7. PMID 25290987
- [Background] Courey MS, Bryant GL Jr, Ossoff RH. Posterior glottic stenosis: a canine model. Ann Otol Rhinol Laryngol. 1998 Oct;107(10 Pt 1):839-46. doi: 10.1177/000348949810701005. PMID 9794612
- [Background] Howard NS, Shiba TL, Pesce JE, Chhetri DK. Photodocumentation of the development of type I posterior glottic stenosis after intubation injury. Case Rep Surg. 2015;2015:504791. doi: 10.1155/2015/504791. Epub 2015 Feb 1. PMID 25705540
- [Background] Lano CF Jr, Duncavage JA, Reinisch L, Ossoff RH, Courey MS, Netterville JL. Laryngotracheal reconstruction in the adult: a ten year experience. Ann Otol Rhinol Laryngol. 1998 Feb;107(2):92-7. doi: 10.1177/000348949810700202. PMID 9486901
- [Background] Colton House J, Noordzij JP, Murgia B, Langmore S. Laryngeal injury from prolonged intubation: a prospective analysis of contributing factors. Laryngoscope. 2011 Mar;121(3):596-600. doi: 10.1002/lary.21403. Epub 2010 Dec 16. PMID 21344442
- [Background] Shinn JR, Kimura KS, Campbell BR, Sun Lowery A, Wootten CT, Garrett CG, Francis DO, Hillel AT, Du L, Casey JD, Ely EW, Gelbard A. Incidence and Outcomes of Acute Laryngeal Injury After Prolonged Mechanical Ventilation. Crit Care Med. 2019 Dec;47(12):1699-1706. doi: 10.1097/CCM.0000000000004015. PMID 31634236
- [Background] Esianor BI, Campbell BR, Casey JD, Du L, Wright A, Steitz B, Semler MW, Gelbard A. Endotracheal Tube Size in Critically Ill Patients. JAMA Otolaryngol Head Neck Surg. 2022 Sep 1;148(9):849-853. doi: 10.1001/jamaoto.2022.1939. PMID 35900743
- [Background] Vahabzadeh-Hagh AM, Marsh-Armstrong BP, Patel SH, Lindenmuth L, Feng Z, Gong R, Lin YA, Pierce T, Loh KJ. Endotracheal tube forces exerted on the larynx and a novel support device to reduce it. Laryngoscope Investig Otolaryngol. 2023 Jul 20;8(4):989-995. doi: 10.1002/lio2.1118. eCollection 2023 Aug. PMID 37621270
- [Background] Bolder PM, Healy TE, Bolder AR, Beatty PC, Kay B. The extra work of breathing through adult endotracheal tubes. Anesth Analg. 1986 Aug;65(8):853-9. PMID 3729022
- [Background] Fiastro JF, Habib MP, Quan SF. Pressure support compensation for inspiratory work due to endotracheal tubes and demand continuous positive airway pressure. Chest. 1988 Mar;93(3):499-505. doi: 10.1378/chest.93.3.499. PMID 3277803
- [Background] Sahn SA, Lakshminarayan S, Petty TL. Weaning from mechanical ventilation. JAMA. 1976 May 17;235(20):2208-12. No abstract available. PMID 946845
- [Background] Southgate MT. Airflow resistances of endotracheal tubes. JAMA. 1977 Mar 28;237(13):1362. doi: 10.1001/jama.237.13.1362a. No abstract available. PMID 576488
- [Background] Behrakis PK, Higgs BD, Baydur A, Zin WA, Milic-Emili J. Respiratory mechanics during halothane anesthesia and anesthesia-paralysis in humans. J Appl Physiol Respir Environ Exerc Physiol. 1983 Oct;55(4):1085-92. doi: 10.1152/jappl.1983.55.4.1085. PMID 6629937
- [Background] Sullivan M, Paliotta J, Saklad M. Endotracheal tube as a factor in measurement of respiratory mechanics. J Appl Physiol. 1976 Oct;41(4):590-2. doi: 10.1152/jappl.1976.41.4.590. PMID 985406
- [Background] Wright PE, Marini JJ, Bernard GR. In vitro versus in vivo comparison of endotracheal tube airflow resistance. Am Rev Respir Dis. 1989 Jul;140(1):10-6. doi: 10.1164/ajrccm/140.1.10. PMID 2751156
- [Background] Shapiro M, Wilson RK, Casar G, Bloom K, Teague RB. Work of breathing through different sized endotracheal tubes. Crit Care Med. 1986 Dec;14(12):1028-31. doi: 10.1097/00003246-198612000-00007. PMID 3780244
- [Background] Orebaugh S, Snyder J. Direct laryngoscopy and endotracheal intubation in adults - UpToDate. Accessed November 22, 2022. https://www.uptodate.com/contents/direct-laryngoscopy-and-endotracheal-intubation-in-adults
- [Background] Farrow S, Farrow C, Soni N. Size matters: choosing the right tracheal tube. Anaesthesia. 2012 Aug;67(8):815-9. doi: 10.1111/j.1365-2044.2012.07250.x. No abstract available. PMID 22775368
- [Background] Brenner MJ, Brodsky MB, Rassekh CH. Reassessing Endotracheal Tube Size in Critically Ill Patients. JAMA Otolaryngol Head Neck Surg. 2023 Feb 1;149(2):188. doi: 10.1001/jamaoto.2022.4273. No abstract available. PMID 36580288
- [Background] Schober P, Schwarte LA, Loer SA. Association Between Endotracheal Tube Size and Outcomes in Critically Ill Patients. JAMA Otolaryngol Head Neck Surg. 2023 Apr 1;149(4):377-378. doi: 10.1001/jamaoto.2022.4995. No abstract available. PMID 36757721